CLINICAL TRIAL: NCT04231162
Title: Effect of an 8-week Bifidobacterium Lactis HN019 Supplementation on Functional Constipation: A Double-blind, Randomized; Placebo-controlled Trial
Brief Title: Effect of an 8-week Bifidobacterium Lactis HN019 Supplementation on Functional Constipation
Acronym: BifidoDigest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH-03643 (PEC18369); 2019-A00720-57 (Other: ID-RCB)
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Functional Constipation
Keywords: Stool frequency; Probiotic; Lactic bacteria; Bifidobacteria; Transit; Quality of life; Constipation symptoms; Diet supplement
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic powder, Bifidobacterium lactis (Experimental)
  Interventions: Dietary Supplement: Active product
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Active product — Bifidobacterium lactis HN019 (probiotic powder). One capsule to consume orally with still water (not sparkling) at room temperature once a day at least 15 minutes before breakfast time.
  Arms: probiotic powder, Bifidobacterium lactis
Dietary Supplement: Control product — Placebo. One capsule to consume orally with still water (not sparkling) at room temperature once a day at least 15 minutes before breakfast time.
  Arms: Placebo

SUMMARY:
This prospective, two-arm (parallel groups), double-blind, randomized, placebo-controlled, multi-center clinical trial will investigate the effects of an 8-week Bifidobacterium lactis HN019 supplementation on stool frequency and on other constipation parameters in adults suffering from functional constipation according to ROME III criteria. The hypothesis is that Bifidobacterium lactis HN019 is superior, in comparison with a placebo, for the increase of stool frequency of at least 1 stool per week.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at visit 1 (D-16)

1. Free-living females and males of age 18 to 70 years (limits included),
2. Body mass index between 18.5 and 34.9 kg/m² (limits included),
3. Meets the ROME III criteria for functional constipation as follows (criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis):

   a. Must meet 2 or more of the following criteria : i. Straining during at least 25% of defecations, ii. Lumpy or hard stools in at least 25% of defecations, iii. Sensation of incomplete evacuation for at least 25% of defecations, iv. Sensation of anorectal obstruction/blockage for at least 25% of defecations, v. Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvis floor), vi. Fewer than three defecations per week, b. Loose stools are rarely present without the use of laxatives, c. Insufficient criteria for Irritable Bowel Syndrome (IBS),
4. Self-reported bowel movement frequency up to 3 stools per week for at least the last 6 months,
5. Participants who agree to maintain their usual level of activity throughout the trial period,
6. Participants who agree to maintain their usual dietary habits and level of exercise etc; i.e. maintain their usual life-style throughout the trial period,
7. Participants who agree not to consume probiotics (except for investigational products), prebiotics, symbiotic, fermented milk, and/or yogurt throughout the trial period,
8. Females of child-bearing potential who agree to use medically approved methods for birth control those including condoms with spermicides, hormonal contraceptives (estrogen and/or progestin products; either oral, intrauterine or epidermal) or intrauterine device with copper. The contraceptive method should have been in place for at least 3 cycles before the beginning of the study, and should not be modified during the study. Postmenopausal women with or without hormone replacement therapy who have been applying the estrogenic or estrogenic/progestin treatment for at least 3 months before the beginning of the study and who agree not to change the treatment during the study,
9. Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects,
10. Consent to participate in the study and willing to comply with the protocol and study restrictions,
11. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to research involving the human person,
12. Participants who agree to be registered on the national file of the volunteers participating in biomedical research.

Inclusion criteria at visit 2 (D-8)

1. Hematological, serum and urine parameters within the normal ranges, or not clinically-relevant. Nonpregnant females, as indicated by negative pregnancy test,
2. 0 to 3 Complete Spontaneous Bowel Movements (CSBM) over the 7 days, per daily diary log between Visit 1 and Visit 2 (Day-15 to Day-9),
3. 100% compliance with placebo consumption over the 7 days, per daily diary log between Visit 1 and Visit 2 (Day-15 to Day-9)
4. 100% completion of daily diary over the 7 days, per daily diary log between Visit 1 and Visit 2 (Day-15 to Day-9).

Inclusion criteria at visit 3 (D0)

1. 0 to 3 CSBMs over the 7 days, per daily diary log between Visit 2 and Visit 3 (Day-7 to Day-1),
2. 100% compliance with placebo consumption over the 7 days, per daily diary log between Visit 2 and Visit 3 (Day-7 to Day-1)
3. 100% completion of daily diary over the 7 days, per daily diary log between Visit 2 and Visit 3 (Day-7 to Day-1).

Exclusion Criteria:

1. Having hypersensitivity or history of allergy to one of the study products,
2. Suffering from a metabolic disorder (diabetes, uncontrolled thyroidal condition) and/or from severe chronic disease (cancer, renal failure, HIV, immunodeficiency, hepatic or biliary disorders, arthritis, uncontrolled cardiac disease) or from a disease found to be inconsistent with the conduct of the study by the investigator,
3. Major gastrointestinal complication (e.g. Crohn's disease, ulcer, IBS-Mixed, IBS-constipation, IBS-Diarrhea, Celiac disease),
4. Lactose-intolerants who consume non-lactose-free dairy products. e.g. regular milk, ice-cream. i.e. Lactose-intolerants who cannot manage their condition (those who manage their intolerance, i.e. who don't consume any product which contain lactose, could be included in the study).
5. Prior abdominal surgery (e.g. gastric by-pass, gastrectomy, gastric band, visceral surgery…) that, in the opinion of the investigator, may present a risk for the participant or confound study results,
6. Current pharmacological treatment related to constipation (e.g., prosecretory agents, antibiotics, antidepressants, antispasmodics, enterokinetic), dietary treatment of constipation (e.g. probiotics, prebiotics, symbiotic, herbal extracts, fibers), or other constipation treatments (e.g. cognitive behavior therapy, acupuncture, biofeedback) or within 1 month before screening,
7. Laxative/suppository use (≥1/month) or laxative/suppository use within 48 hours of screening (rescue medications - e.g., laxatives, suppositories and rescue procedures- e.g., enemas, allowed for intolerable symptoms during study),
8. Daily consumption of probiotics, prebiotics, symbiotic, fermented milk, and/or yogurt containing probiotics within 2 weeks prior to screening,
9. Use of any drug or dietary supplement during at least 7 consecutive days known to cause constipation (e.g. iron, opioids, sucralfate, misoprostol, 5-HT#-antagonists, antacids with magnesium, calcium or aluminium, antidiarrheal medication, anticholinergic agents, calcium supplements, calcium channel blockers, tricyclic antidepressants or NSAIDs) within 1 month before screening,
10. Clinically significant underlying systemic illness that may preclude the participant's ability to complete the trial or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness),
11. Systemic steroid use within 1 month before screening,
12. Eating disorder (e.g., anorexia, bulimia, etc.),
13. Having a lifestyle deemed incompatible with the study according to the investigator e.g., specific diet (vegetarian, vegan, hypocaloric), intense physical activity > 10 hours / week, etc,
14. Self-declare history of alcohol abuse (for females: >3 drinks on any single day and >7 drinks per week; for males: >4 drinks on any single day and >14 drinks per week),
15. Self-declare use of illicit drugs,
16. Pregnant or lactating female, or pregnancy planned during study period,
17. Planning to travel for a long time during the study duration or not able to be contacted for emergency reason during the study,
18. Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study,
19. Presenting a psychological or linguistic incapacity to understand and sign the informed consent,
20. Participating in another clinical trial or in exclusion period from a previous clinical trial,
21. Participants under administrative or legal supervision,
22. Participants who would receive more than 4500 euros as indemnities for their participation in clinical trial within the 12 last months, including the indemnities for the present study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline of stool frequency | Baseline (Day-15 to Day-9 and Day-7 to Day-1) and Intervention (Day1 to Day28 and Day30 to Day57)
  Complete Spontaneous Bowel movement / week (reported in daily diaries)

SECONDARY OUTCOMES:
Stool consistency | Baseline (Day-15 to Day-9 and Day-7 to Day-1) and Intervention (Day1 to Day28 and Day30 to Day57)
  For each stool by using the Bristol Stool Scale. classify the form of human faeces into seven categories: ypes 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 tending towards diarrhoea, and 6 and 7 indicate diarrhoea
Degree of straining | Baseline (Day-15 to Day-9 and Day-7 to Day-1) and Intervention (Day 1 to Day 28 and Day 30 to D57)
  For each stool by using Visual analogue scale, a 100 mm long horizontal VAS, anchored at 0 mm (not at all), 25 mm (a little bit), 50 mm (a moderate amount), 75 mm (a great deal) and 100 mm (an extreme amount).
Abdominal pain severity | Baseline (Day-15 to Day-9 and Day-7 to Day-1) and Intervention (Day1 to Day28 and Day30 to Day57)
  For each stool by using Visual analogue scale, rated using a 100 mm long horizontal VAS, anchored at 0 mm (none), 25 mm (mild), 50 mm (moderate), 75 mm (severe) and 100 mm (very severe).
Bloating severity | Baseline (Day-15 to Day-9 and Day-7 to Day-1) and Intervention (Day1 to Day28 and Day30 to Day57)
  For each stool by using Visual analogue scale, rated using a 100 mm long horizontal VAS, anchored at 0 mm (none), 25 mm (mild), 50 mm (moderate), 75 mm (severe) and 100 mm (very severe).
Constipation symptoms assessment by the participant | Day 0 (baseline, Visit 3), Day 29 (Visit 4, 4 weeks) and Day 58 (Visit 5, 8 weeks)
  Patient Assessment of Constipation SYMptoms (PAC-SYM) questionnaire: global score, abdominal symptoms, rectal symptoms and symptoms associated to stool, measures the severity of constipation symptoms over the past 2 weeks; no symptom, 0; mild, 1;moderate, 2. severe, 3; very severe, 4
Quality of life related to constipation assessment by the participant | Day 0 (baseline, Visit 3), Day 29 (Visit 4, 4 weeks) and Day 58 (Visit 5, 8 weeks)
  Patient Assessment Constipation Quality Of Life (PAC-QOL) 28-question survey. The questions are comprised of four subscales (worries and concerns, physical discomfort, psychosocial discomfort, and satisfaction) and an overall scale. Not at all, 0; A little bit, 1; Moderately, 2; Quite a bit, 3; Extremely, 4
Use of rescue medication | Day 0 (baseline, Visit 3), Day 29 (Visit 4, 4 weeks) and Day 58 (Visit 5, 8 weeks)
  Need and use of rescue medication (laxative) during the study (reported in daily diaries)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Metreau, MD, Principal Investigator — BioFortis
Locations (4):
- France (4):
  - CEN, Dijon
  - Eurofins Optimed, Gières
  - Institut Pasteur de Lille, Lille
  - Biofortis, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ala-Jaakkola R, Forssten SD, Cheng J, Griffon F, Metreau I, Sturm Y, Lecerf JM, Donazzolo Y, Junnila J, Nordlund A, Hibberd A, Ouwehand AC, Ibarra A. Effect of an 8-Week Bifidobacterium lactis HN019 Supplementation on Functional Constipation: A Multi-Center, Triple-Blind, Randomized, Placebo-Controlled Trial. Mol Nutr Food Res. 2025 Sep;69(17):e70081. doi: 10.1002/mnfr.70081. Epub 2025 May 5. PMID 40320938